CLINICAL TRIAL: NCT07145164
Title: Interleukin-15 to Promote Post-ART Control of HIV
Acronym: INTERRUPT-HIV
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Peluso, MD (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor-Investigator, Michael Peluso, MD, Assistant Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-44404
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: HIV; IL-15; N-803; Anktiva
MeSH Terms: interventions — ALT-803

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-803 (Experimental): Participants in this arm will receive the active study drug during the blinded portion (Phase A) of the trial. They will receive the active study drug during the open-label portion (Phase B) of the trial.
  Interventions: Drug: N-803
- Placebo (Placebo Comparator): Participants in this arm will receive placebo during the blinded portion (Phase A) of the trial. They will receive the active study drug during the open-label portion (Phase B) of the trial.
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: N-803 — This is the active drug.
  Arms: N-803
Drug: Saline placebo — This is the placebo.
  Arms: Placebo

SUMMARY:
Even though HIV medicine stops the virus from making more copies of itself, the virus remains in the body by hiding inside of immune cells. This hidden virus is referred to as the "latent reservoir." Researchers on this team are studying whether stimulating the immune system can change the nature of the latent reservoir and if this could help people control HIV without the need to take regular HIV medicine.

This study is testing a drug called N-803. N-803 is also known as Interleukin-15 or "IL-15", a powerful and long lasting protein that can affect the immune system by stimulating immune cells such as CD8+ T cells and natural killer (NK) cells. CD8+ T cells and NK cells are both crucial for eliminating infected cells. The drug is FDA-approved for the treatment of bladder cancer, but in this study the drug is being used experimentally for HIV.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 and ≤ 70 years at the time of screening
* Documented HIV-1 infection
* On continuous ART for at least 6 months without any interruptions of greater than 14 consecutive days within the preceding 6 months
* Plasma HIV RNA levels less than 200 copies/mL at each determination in the previous 6 months
* Screening CD4+ T-cell count ≥ 350 cells/mm3
* Willingness to interrupt ART as part of the study transient treatment interruption

Exclusion Criteria:

* On an ART regimen that includes a non-nucleoside reverse transcriptase inhibitor, unable to switch to a different regimen
* Receipt of any long-acting ART medication (e.g., injectable cabotegravir/rilpivirine, lenacapavir) in the two years preceding screening.
* Known resistance to two or more classes of ART drugs and/or the inability to construct another fully suppressive regimen
* Evidence of HIV "elite" control immediately prior to ART initiation
* Screening platelets < 125,000/mm3
* Screening hemoglobin < 12.5 g/dL for men and <11.5 for women
* History of an AIDS-defining illness according to CDC criteria
* History of HIV-associated malignancy
* Non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the 36 months preceding screening, or for whom such therapies are expected in the subsequent 12 months.
* Active Hepatitis B (Hep B) infection (defined as Hep B surface antigen (sAg) positive or HBV DNA positive)
* Active Hepatitis C (Hep C) infection (defined as Hep C Ab positive or indeterminate with detectable Hep C RNA)
* Chronic liver disease
* Chronic kidney disease
* Active and poorly controlled atherosclerotic cardiovascular disease
* QTc interval >450msec (male) or >470msec (female)
* Pregnant, breastfeeding, or unwilling to use contraception to prevent pregnancy during participation in the study and until 6 months resumption of ART
* Unable or unwilling to use barrier protection or pre-exposure prophylaxis (PrEP) in the partner, with sexual partners not known to have HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Solicited Adverse Events | Within 7 days after dosing.
  Frequency and grade of each solicited systemic reactogenicity AE (malaise, participant-measured body temperature, fatigue, headache, chills, nausea, muscle aches/pain, joint pain).
Safety - Unsolicited Adverse Events | Within 7 days after dosing.
  Frequency and grade of unsolicited AEs.

SECONDARY OUTCOMES:
Time to Rebound | 52 weeks after treatment interruption.
  Difference in time-to-viral rebound, defined as the first of two consecutive viral loads > the limit of quantification of the assay, between those who previously received the intervention and those who previously received placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set with longitudinal clinical data will be shared upon the publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code